CLINICAL TRIAL: NCT03230747
Title: Early Feasibility Study of the Edwards SAPIEN M3 System for the Treatment of Mitral Regurgitation
Brief Title: SAPIEN M3 EFS: Early Feasibility Study of the Edwards SAPIEN M3 System for the Treatment of Mitral Regurgitation
Acronym: SAPIEN M3 EFS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2017-03
Record Dates: First submitted 2017-07-24; First posted 2017-07-26 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Mitral Regurgitation; Mitral Disease
Keywords: Transcatheter Mitral Valve Replacement; SAPIEN M3
MeSH Terms: conditions — Mitral Valve Insufficiency; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- TMVR (Experimental): Subjects will undergo transcatheter mitral valve replacement
  Interventions: Device: Edwards SAPIEN M3 System

INTERVENTIONS:
Device: Edwards SAPIEN M3 System — SAPIEN M3 System includes the SAPIEN M3 valve and the SAPIEN M3 dock

SUMMARY:
This study will evaluate the safety and functionality of the SAPIEN M3 System in patients with symptomatic, severe MR and will provide guidance for future clinical study designs utilizing the SAPIEN M3 System.

DETAILED DESCRIPTION:
Prospective, single-arm, multicenter early feasibility study

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. MR ≥ 3+
3. NYHA functional class ≥ II
4. High risk of cardiovascular surgery
5. Hemodynamically stable while on heart failure medication for at least 2 weeks before the procedure
6. The study patient has been informed of the nature of the study, agrees to its provisions and has provided written informed consent.

Exclusion Criteria:

1. Mitral anatomy that would preclude appropriate delivery and deployment of the dock or valve
2. Cardiac imaging evidence of intracardiac mass, thrombus or vegetation
3. Significant risk of LVOT obstruction
4. Severe right ventricular dysfunction
5. LV Ejection Fraction <30%
6. Patient is inoperable
7. Prior surgical or interventional treatment of mitral valve preventing appropriate device access and deployment
8. Need for aortic, tricuspid or pulmonic valve replacement
9. Presence of mechanical aortic valve prosthesis
10. History of cardiac transplantation
11. History of recurrent and/or unprovoked deep vein thrombosis or pulmonary embolism
12. Clinically significant untreated coronary artery disease requiring revascularization
13. Any percutaneous cardiovascular intervention, cardiovascular surgery, or carotid surgery within 30 days.
14. Stroke or transient ischemic attack within 90 days of the procedure
15. Myocardial infarction within 30 days of the procedure
16. Active bacterial endocarditis within 180 days of the procedure
17. Inability to tolerate or a medical condition precluding treatment with anti-thrombotic therapy
18. Leukopenia, anemia, thrombocytopenia, history of bleeding diathesis or coagulopathy, or hypercoagulable states
19. Hospitalization for CHF or hemodynamic instability requiring inotropic support or intra-aortic balloon pump within 30 days.
20. Irreversible, severe pulmonary hypertension
21. Patients with renal insufficiency or receiving renal replacement therapy
22. Liver disease or significantly abnormal liver function test results
23. Refusal of blood products
24. Female who is pregnant or lactating
25. Estimated life expectancy < 12 months
26. Participating in another investigational drug or device study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2021-06-16 (Actual); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Technical Success | At the end of the procedure
  Defined as meeting all the following:
  * Alive
  * Successful access, delivery and retrieval of the delivery systems
  * Deployment of the devices in the intended position
  * Freedom from emergency surgery or reintervention related to the device or access procedure

SECONDARY OUTCOMES:
Reduction in mitral regurgitation (MR) | 30 Days
  Reduction in MR to 0 or 1+

CONTACTS AND LOCATIONS:
Locations (9):
- United States (8):
  - Cedars-Sinai Medical Center Heart Institute, Los Angeles, California
  - California Pacific Medical Center, San Francisco, California
  - Emory University, Atlanta, Georgia
  - Evanston/ Northshore University, Evanston, Illinois
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Intermountain Medical Center, Murray, Utah
  - Sentara Cardiovascular Research Institution, Norfolk, Virginia
- St. Paul's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No